CLINICAL TRIAL: NCT03616886
Title: A Phase I/II Study of Paclitaxel Plus Carboplatin and Durvalumab (MEDI4736) With or Without Oleclumab (MEDI9447) for Previously Untreated Locally Recurrent Inoperable or Metastatic Triple-negative Breast Cancer
Brief Title: Paclitaxel + Carboplatin + Durvalumab With or Without Oleclumab for Previously Untreated Locally Recurrent Inoperable or Metastatic TNBC
Acronym: SYNERGY
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IJB-SYNERGY-012017
Record Dates: First submitted 2018-07-16; First posted 2018-08-06 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Triple Negative Breast Cancer
Keywords: Breast cancer; Triple negative; Metastatic; Previously untreated; Locally Recurrent Inoperable
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Neoplasm Metastasis | interventions — Paclitaxel; Carboplatin; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase I and Phase II Arm A (Experimental): Patients are treated with paclitaxel, carboplatin, durvalumab and oleclumab.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: MEDI4736; Drug: MEDI9447
- Phase II Arm B (Active Comparator): Patients are treated with paclitaxel, carboplatin and durvalumab.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: MEDI4736

INTERVENTIONS:
Drug: Paclitaxel — Patients will be randomized between chemotherapy (paclitaxel and carboplatin) with immunotherapy including durvalumab with or without oleclumab (1:1 ratio).
Drug: Carboplatin — Patients will be randomized between chemotherapy (paclitaxel and carboplatin) with immunotherapy including durvalumab with or without oleclumab (1:1 ratio).
Drug: MEDI4736 — Patients will be randomized between chemotherapy (paclitaxel and carboplatin) with immunotherapy including durvalumab with or without oleclumab (1:1 ratio).
  Other Names: Durvalumab
Drug: MEDI9447 — Patients will be randomized between chemotherapy (paclitaxel and carboplatin) with immunotherapy including durvalumab with or without oleclumab (1:1 ratio).
  Other Names: Oleclumab
  Arms: Phase I and Phase II Arm A

SUMMARY:
The combination of chemotherapy with PD-1 immune checkpoint blockade agents demonstrated promising results especially in the neo-adjuvant and early metastatic setting in TNBC. However, a substantial proportion of patients do not derive benefit from this approach.

CD73 is an adenosine-generating enzyme overexpressed in several cancers and associated with poor prognosis and reduced anti-tumor immunity in TNBC. Monoclonal antibodies directed against CD73 could help to reprogram the tumor microenvironement by decreasing the adenosine mediated immunosuppression, particularly as a synergistic immunotherapeutic combination with immune checkpoint blockade.

The SYNERGY trial investigates the role of an anti-CD73 (MEDI9447) in a randomized phase II trial evaluating the efficacy and safety of the combination of chemotherapy (paclitaxel + carboplatin) with immunotherapy (durvalumab [anti-PD-L1] +/- MEDI9447 [anti-CD73]) in previously untreated locally recurrent inoperable or metastatic TNBC.

A large translational research program is planned including baseline and dynamic biomarkers

DETAILED DESCRIPTION:
The trial consists of two parts:

PHASE I Part 1 is a phase I trial examining the combination of paclitaxel, carboplatin, durvalumab and oleclumab in order to define the recommended phase II dose (RP2D) of oleclumab in this treatment combination.

The period for DLT evaluation is defined as the time from receiving the first dose of oleclumab until the planned administration of the third dose; this corresponds to 28 days after receiving the first dose of oleclumab in case no treatment interruption occured.

Patients who develop a DLT will stop study treatment permanently.

PHASE II Part 2 is a multicenter, randomized, open-label trial investigating the role of an anti-CD73 monoclonal antibody (oleclumab) in combination with an anti-PD-L1 antibody (durvalumab) plus chemotherapy (paclitaxel + carboplatin) as first-line treatment for locally recurrent inoperable or metastatic TNBC.

Patients will be randomized between chemotherapy (paclitaxel and carboplatin) with immunotherapy including durvalumab with or without oleclumab (1:1 ratio).

PHASE I and PHASE II

Paclitaxel and carboplatin will be given weekly for a total of 12 injections. Immunotherapy (durvalumab with or without oleclumab) will be given as long as the patient benefits. Premature discontinuation of paclitaxel/carboplatin or discontinuation of durvalumab/oleclumab is indicated in case of:

* Progressive disease (PD) using RECIST v1.1 criteria or iRECIST assessed locally
* Unacceptable toxicity
* Intercurrent illness that necessitates discontinuation of study treatment
* Investigator's decision to withdraw the subject
* Pregnancy
* Subject noncompliance with the study treatment or procedure requirements
* Withdrawal of consent to treatment
* Death
* Administrative reasons requiring cessation of study treatment.

Initial disease status will be evaluated by imaging studies (contrast-enhanced CT scan of the chest, the abdomen and the pelvis or MRI of the chest, the abdomen and the pelvis) during the screening phase. Disease status will be followed by imaging studies at weeks 8 (± 3 days), 16 (± 3 days) and 24 (± 3 days) post start of treatment (allowing efficacy data to be captured as close to 24 weeks post start of study treatment as possible for a more accurate evaluation of DCR). Thereafter imaging will continue every 12 weeks (± 3 days; contrast-enhanced CT scan or MRI) independent of any treatment delays.

Patients who stopped all study treatments for reasons other than PD will continue post-treatment imaging studies for disease status follow-up as described in the schedule of assessment until verified PD, start of a new anti-cancer treatment, withdrawal of consent to study participation, death, or end of the study whichever comes first.

Note: Pseudo-progression related to immunotherapy: Patients experiencing PD as defined by RECIST v1.1 can continue the study treatment in case of good clinical condition assessed by a stable or even improved ECOG performance status. If the next assessment of tumour burden (8 weeks later) confirms PD (as defined by iRECIST) study treatment must be discontinued. Unconfirmed PD as defined by iRECIST (iUPD) can only be assigned for the first 2 imaging assessments (week 8 and week 16) and several times as long as confirmed progression (iCPD) is not confirmed at the next assessment. If PD is not confirmed, reassessments continue as originally planned.

ELIGIBILITY:
Inclusion Criteria:

1. Age of ≥ 18 years
2. Female
3. Life expectancy of a least 12 weeks
4. Body weight above 35kg
5. The locally recurrent or metastatic relapse must be histologically confirmed TNBC in patients not previously treated with systemic treatment and which cannot be treated with curative intent. Newly diagnosed patients with de-novo metastatic disease are eligible
6. Estrogen receptor (ER) and progesterone receptor (PR) negativity (< 1% positive staining cells in the invasive tumour) determined locally using IHC per ASCO/CAP criteria
7. Human epidermal growth factor receptor 2 (HER2) negativity (negative IHC staining [score 0 or 1] or negative fluorescence in situ hybridization [FISH] based on the ASCO/CAP guidelines and recommendations) and determined locally59 Note: patients initially diagnosed with hormone receptor-positive and/or HER2-positive breast cancer OR de novo metastatic patients with a primary tumor hormone receptor-positive (weak positivity or ER negativity and PR positivity) considered as non-clinically relevant are eligible if the tumor biopsy obtained from a local recurrence or distant metastasis site confirms the TNBC disease.
8. Confirmed tumour PD-L1 and CD73 IHC assessment as documented through central testing of a representative tumour tissue specimen for stratification purposes (only for phase II)
9. Provision of recurrence/metastatic tissue samples from resections, core-needle biopsies or excisional, incisional, punch, or forceps biopsies:

   * at least 1 FFPE [Formalin-Fixed paraffin-embedded] tumour tissue and 1 frozen core as a priority, if feasible 2 additional fresh tumour tissue cores should be collected too)
   * Fine-needle aspiration (FNA) (defined as samples that do not preserve tissue architecture and yield cell suspension and/or smears), brushing, and cell pellets from cytology samples are not acceptable.

   Note 1: If the patient has just performed a metastatic lesion biopsy, she is eligible only if an archived FFPE tissue sample (or at least 20 unstained slides, freshly cut for the purposes of the study) of the metastatic lesion is available. In this situation only, frozen/fresh cores are not mandatory.

   Note 2: In case of a de-novo metastatic disease, if a biopsy of a metastatic lesion is not feasible, the patient is eligible if a biopsy of the primary lesion is available.
10. Provision of an archived FFPE diagnostic biopsy or surgical primary breast tumour sample (or at least 20 unstained slides, freshly cut for the purposes of the study).

    Note: In case of neoadjuvant treatment (before surgery), the diagnostic biopsy is preferable.
11. At least 6 months elapsed between the completion of treatment with curative intent (e.g., the date of primary breast tumour surgery or the date of last adjuvant chemotherapy administration, whichever occurred last) and first documented local or distant disease recurrence (NOTE: not applicable for de-novo metastatic disease)
12. At least one measurable disease based on RECIST v1.1. Tumour lesions in a previously irradiated area are considered measurable, if progression has been demonstrated in such lesions
13. Adequate organ function:

    1. Absolute neutrophil count (ANC) ≥ 1500/μl (without the addition of growth factors)
    2. Platelets [PLT] ≥ 100000/μl (without the addition of growth factors/prior transfusions)
    3. Hemoglobin (Hb) ≥ 10 g/dl (without the addition of growth factors/prior transfusions)
    4. Creatinine ≤ 1.5 x upper limit of normal (ULN) OR estimated glomerular filtration rate (eGFR) ≥ 60 ml/min as calculated using the method standard for the institution. If eGFR is lower than 60 ml/min, a 24-hour urine creatinine clearance can be performed to rule out an underestimation of the eGFR.
    5. Total serum bilirubin (TBL) ≤ 1.5 x ULN unless the subject has documented Gilbert syndrome in which case up to 3 x ULN is acceptable
    6. Aspartate and alanine aminotransferase (AST/ALT) ≤ 2.5 x ULN unless liver metastases are present, in which case it must be ≤ 5 x ULN
    7. International Normalized Ratio (INR) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as INR and activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants
14. Performance status (PS) of 0 or 1 on the ECOG Performance scale
15. Female subjects of childbearing potential (FSCP) must be willing to use one highly effective method of contraception (detailed at protocol section 6.6.) for the course of the study through 6 months after the last study drug administration. FSCP must have a negative serum pregnancy test done within the 28 days before treatment start. FSCP are those who have not been surgically sterilized or have not been free of menses for at least 1 year.
16. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
17. Absence of any concurrent illness that would preclude the evaluation of safety
18. Agreement to provide tissue and blood samples for research purposes
19. Written informed consent must be given according to ICH/GCP, and national/local regulations before patient enrolment
20. Applicable to France only: Affiliated to the French Social Security System

Exclusion Criteria:

1. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   1. Patients with vitiligo or alopecia
   2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   3. Any chronic skin condition that does not require systemic therapy
   4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   5. Patients with celiac disease controlled by diet alone
2. Current or prior treatment with immunosuppressive medication within 14 days prior to enrolment. The following are exceptions to this criterion:

   1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
   2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
   3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication
3. Any live, attenuated vaccine administered within 28 days prior to enrolment or anticipation that such a live attenuated vaccine will be required during the study
4. Chronic daily treatment with non-steroidal anti-inflammatory drug (NSAID) (occasional use for the symptomatic relief of medical conditions, for example, headache, fever is allowed)
5. Active infection including

   1. Tuberculosis (TB) (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice)
   2. Hepatitis B (known positive HBV surface antigen (HBsAg) result). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible.
   3. Hepatitis C. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
   4. Human immunodeficiency virus (positive HIV 1/2 antibodies).
6. Treatment with systemic immunostimulatory agents, including but not limited to, interferon (IFN)-alpha, IFN-beta, interleukin (IL)-2, conjugated IL-2 cytokines within 42 days or five half-lives of the drug, whichever is longer, prior to screening
7. Previous treatment with immune checkpoint inhibitors (e.g. anti-PD-1, anti-PD-L1 including durvalumab, anti-Cytotoxic T-lymphocyte-associated molecule-4), anti-CD73 antibodies, adenosine A2A receptor antagonists, or prior treatment with CD137 agonists/OX-40 agonists or any other antibody or drug targeting T-cell co-stimulation or other immunomodulatory therapies
8. Any unresolved toxicity NCI CTCAE Grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo and the laboratory values defined in the inclusion criteria
9. Known hypersensitivity reactions to the study drugs or to any of the excipients, premedications (acetaminophen/paracetamol, diphenhydramine or equivalent antihistamine and methylprednisolone or equivalent glucocorticoid) and to other platinum containing compounds
10. Untreated central nervous system (CNS) metastases and/or carcinomatous meningitis.

    Subjects with previously treated brain metastases with local treatment (stereotactic radiosurgery or whole brain radiation therapy) may participate provided they have stable brain metastases on a recent brain MRI (performed during the 2 weeks prior inclusion) and have measurable disease outside the CNS.

    Note: Known brain metastases are considered active (and not eligible for trial), if any of the following criteria are applicable:
    1. Recent brain imaging demonstrates progression of existing and/or appearance of new lesions
    2. Neurological symptoms attributed to brain metastases have not returned to baseline
    3. Steroids were used for management of symptoms related to brain metastases within 14 days of enrolment
    4. Completion of local therapy for brain metastases within 28 days of enrolment
11. Major surgical procedure (as defined by the principal investigator) within 28 days prior to enrolment. Note: Local surgery of isolated lesions for palliative intent is acceptable.
12. Uncontrolled intercurrent illness, including but not limited to,

    1. Symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia. Patients previously treated with anthracyclines are eligible if a recent cardiac work up (< 6 months) demonstrated a normal left ventricular ejection fraction (LVEF≥50%).
    2. Interstitial lung disease
    3. Serious chronic gastrointestinal conditions associated with diarrhoea
    4. Psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
13. Past medical conditions, including,

    1. Class II-IV congestive heart failure
    2. Myocardial infarction within 12 months prior enrolment,
    3. Deep vein thrombosis (DVT) or thrombo-embolic event within 12 months prior to enrolment
    4. History of stroke or transient ischemic attack requiring medical therapy
    5. Intra-abdominal inflammatory process within the last 12 months prior to enrolment such as, but not limited to, diverticulitis, peptic ulcer disease, or colitis
    6. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g. bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis
    7. History of another primary malignancy except for malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence, adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease, adequately treated carcinoma in situ without evidence of disease
    8. Status post allogeneic bone marrow transplantation or solid organ transplantation
14. Pregnant or lactating women.
15. Applicable to France only: Vulnerable persons according to the article L.1121-6 of the Public Health Code, adults who are the subjects of a measure of legal protection or unable to express their consent according to article L.1121-8 of the Public Health Code

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase I:The adverse events (AEs) | Through the Phase I, approximately 7 months
  Safety and tolerability will be assessed by monitoring frequency, duration and severity of adverse events (AEs).
Phase II: Clinical Benefit of oleclumab in combination with chemotherapy and durvalumab by the comparing the CB rate at 24 weeks from the 1st dose of study drug administration between patients treated with or without the anti-CD73 antibody oleclumab | At 24 weeks from the 1st study drug administration
  CB is defined as a patient who achieved CR or PR or demonstrated SD at 24 weeks from the 1st dose of study drug administration based on RECIST v1.1.

SECONDARY OUTCOMES:
Phase I: Recommended phase II dose (RP2D) of oleclumab in combination with chemotherapy and durvalumab | through study completion, approximately 50 months
  Safety and tolerability will be assessed by monitoring frequency, duration and severity of adverse events (AEs) including Dose limiting toxicities (DLTs) as defined per protocol.
Phase II: Efficacy of oleclumab in combination with chemotherapy and durvalumab by comparing the OR rate (ORR; CR + PR) and the duration of response (DOR) between patients treated with or without the anti-CD73 antibody oleclumab. | through study completion, approximately 50 months
  OR is defined as a patient (in the intent-to treat population) who achieved a CR or PR as best overall response (BOR) based on RECIST v1.1.
Phase II: Efficacy of oleclumab in combination with chemotherapy and durvalumab by comparing the OR rate (ORR; CR + PR) and the duration of response (DOR) between patients treated with or without the anti-CD73 antibody oleclumab. | through study completion, approximately 50 months
  DOR is defined as the time from documentation of first tumour response to disease progression based on RECIST v1.1.
Phase II: the progression-free survival (PFS) | through study completion, approximately 50 months
  PFS is defined as the time from 1st study drug administration to the first documented disease progression based on RECIST v1.1 or death due to any cause, whichever occurs first. (Subjects who are alive and progression free at the time of analysis will be censored at the time-point of their last tumour assessment by imaging.)
Phase II: overall survival (OS) | through study completion, approximately 50 months
  OS is defined as the time from 1st study drug administration to death due to any cause. (Subject without documented death at the time of the analysis will be censored at the date of the last follow-up.)
Phase II: AEs assessment based on CTCAE 5.0. | through study completion, approximately 50 months
  Frequency, duration and severity of AEs assessment based on CTCAE 5.0.
Phase II: Efficacy, clinical and survival benefits of oleclumab in combination with chemotherapy and durvalumab according to PD-L1 and CD73 expression. | through study completion, approximately 50 months
  PD-L1 and CD73 expression will be assessed using immunohistochemistry (IHC) on the screening FFPE tumour tissue lesion biopsy by a central laboratory prior to randomization for stratification purposes

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Buisseret, Study Chair — Jules Bordet Institute
Locations (16):
- Belgium (7):
  - Institut Jules Bordet, Brussels
  - Cliniques universitaires Saint Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - UZ Leuven Gasthuisberg, Leuven
  - CHU UCL Namur Sainte-Elisabeth, Namur
  - Clinique St Pierre, Ottignies
  - Sint-Augustinus, GZA Ziekenhuizen, Wilrijk
- France (9):
  - CHU Besançon, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Institut Paoli-Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - CHU Poitiers, Poitiers
  - Centre Henri Becquerel, Rouen
  - Hôpitaux Universitaires de Strasbourg, Strasbourg